CLINICAL TRIAL: NCT02485652
Title: A Single Arm, Open-label, Phase 2 Study Evaluating the Efficacy, Safety and PK of HM61713 in Patients With T790M-positive NSCLC After Treatment With an Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor
Brief Title: Phase II Trial of HM61713 for the Treatment of ≥2nd Line T790M Mutation Positive Adenocarcinoma of the Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study termination by the Sponsor
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMSI-202; 2015-001435-21 (EudraCT Number)
Record Dates: First submitted 2015-06-22; First posted 2015-06-30 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; EGFR-TKI; non small cell lung cancer; HM61713; T790M-positive; lung cancer; Phase II; Olmutinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — olmutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HM61713 (Experimental): HM61713 800 mg (2 x 400 mg tablets) once daily (QD)
  Interventions: Drug: HM61713

INTERVENTIONS:
Drug: HM61713 — 800 mg QD continuously in 21-day cycles until disease progression determined by investigator assessment per RECIST version 1.1, and as long as, in the investigator"s opinion, they are benefiting from study treatment and they do not meet any of treatment discontinuation criteria.
  Other Names: Olmutinib

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of HM61713 in patients with T790M-positive non-small cell lung cancer (NSCLC) after treatment with an epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI).

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase 2 study to assess the anti-tumor efficacy of oral single agent HM61713 administered to patients with T790M-positive NSCLC after treatment with an EGFR-TKI as measured by objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 20 years of age
* Cytologically or histologically confirmed adenocarcinoma of locally advanced or metastatic NSCLC which is not amenable to curative surgery or radiotherapy
* Radiologically confirmed disease progression after at least one line of treatment with an EGFR-TKI
* At least one documented EGFR mutation which is known to be related with susceptibility to EGFR-TKIs (including G719X, exon 19 deletion, L858R, and L861Q)
* World Health Organization (WHO) performance score of 0 to 1 with life expectancy of at least 3 months
* Centrally confirmed T790M mutation positive tumor status from a tumor sample taken after confirmation of disease progression on the most recent anticancer treatment regimen
* At least one lesion (excluding the brain), not previously irradiated that can be accurately measured per RECIST version 1.1
* Adequate hematological and biological function
* Females of child-bearing potential must agree to use adequate contraception and for 3 months after the last dose of study drug
* Male patients should be documented to be sterile or agree to use barrier contraception
* Recovery to ≤ Grade 1 or baseline of any toxicities, except for stable sensory neuropathy ≤ Grade 2 and alopecia

Exclusion Criteria:

* Known history of hypersensitivity to active or inactive excipients of HM61713 or drugs with a similar chemical structure of HM61713
* Previous treatment with anticancer therapies, EGFR-TKI, HM61713, or other drugs that target T790M-positive mutant EGFR with sparing of wild-type, investigational agent(s) within 28 days prior to the first administration of study drug, radiotherapy
* Any non-study related significant surgical procedures within the past 28 days prior to the first administration of study drug
* Spinal cord compression, leptomeningeal carcinomatosis or active symptomatic brain metastases
* History of any other malignancy
* Clinically significant uncontrolled condition(s)
* Active or chronic pancreatitis
* Anyone with cardiac abnormalities or history
* Presence or history of ILD, drug-induced ILD, or presence of radiation pneumonitis
* Pregnant or breast feeding
* In the opinion of the investigator, the patient is an unsuitable candidate to receive HM61713

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess the anti-tumor efficacy of HM61713 as measured by objective response rate (ORR).

SECONDARY OUTCOMES:
Disease control rate (DCR), defined as the proportion of patients with a documented CR, PR, and SD during the treatment cycles according to the RECIST version 1.1 | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess clinical efficacy of HM61713 regarding disease control rate (DCR).
Duration of overall tumor response (DR), defined as the interval between the date of the first observation of tumor response (CR or PR) and the date of disease progression or death | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess clinical efficacy of HM61713 regarding Duration of overall tumor response (DR).
Progression-free survival (PFS), defined as the time from first administration of study drug to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess clinical efficacy of HM61713 regarding Progression-free survival (PFS).
Overall survival (OS), defined as the time from first administration of study drug until death from any cause | From first dose to end of study or date of death from any cause whichever came first, assessed up to 48 months
  To assess clinical efficacy of HM61713 regarding Overall survival (OS).
Time to progression (TTP), defined as the time from first administration of study drug to determination of tumor progression by RECIST version 1.1 | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess clinical efficacy of HM61713 regarding Time to progression (TTP).
Tumor shrinkage calculated as absolute change and percentage change from baseline in sum of tumor size at each assessment using RECIST tumor response | At baseline and every 6 weeks from time of first dose until date of progression, assessed up to 12 months
  To assess clinical efficacy of HM61713 regarding tumor shrinkage.
Peak concentration (Cmax) of HM61713 | Pre-dose (-30 to 0 mins) and 1 hour (± 5 mins), 3, 4, 6 hours (± 10 mins) on Day 1 and Day 15 of Cycle 1 and pre-dose (-30 to 0 mins) only on Day 8 of Cycle 1 and Day 1 of Cycle 2 (Day 22)
  To determine the pharmacokinetic (PK) profile of HM61713.
Trough plasma concentration (Ctrough) of HM61713 | Pre-dose (-30 to 0 mins) and 1 hour (± 5 mins), 3, 4, 6 hours (± 10 mins) on Day 1 and Day 15 of Cycle 1 and pre-dose (-30 to 0 mins) only on Day 8 of Cycle 1 and Day 1 of Cycle 2 (Day 22)
  To determine the pharmacokinetic (PK) profile of HM61713.
Area under the plasma concentration time curve over the 24-hour dosing interval (AUC) of HM61713 | Pre-dose (-30 to 0 mins) and 1 hour (± 5 mins), 3, 4, 6 hours (± 10 mins) on Day 1 and Day 15 of Cycle 1 and pre-dose (-30 to 0 mins) only on Day 8 of Cycle 1 and Day 1 of Cycle 2 (Day 22)
  To determine the pharmacokinetic (PK) profile of HM61713.
Patient reported outcomes (PROs) | At baseline and every 6 weeks from time of discontinuation, assessed up to 24 months
  To assess patient reported outcomes (PROs) of health-related quality of life (HRQoL), disease/treatment-related symptoms of lung cancer, and general health status.
ECG/QTc (absolute values and change from baseline) | Adverse events will be collected from baseline until 28 days after the last dose
  To evaluate the effect of HM61713 on the QT interval.
Incidence of reported AEs and abnormal laboratory tests (AEs will be assessed using the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4). | Adverse events will be collected from baseline until 28 days after the last dose
  To assess the safety and tolerability of HM61713.
QTc interval as assessed by digital ECG with central reading. The QT interval will be rate-corrected using 3 methods: QTcF, QTcB and QTcS. | Adverse events will be collected from baseline until 28 days after the last dose
  To assess the safety and tolerability of HM61713.

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, M.D., Ph.D, Principal Investigator — Sungkyunkwan University, Samsung Medical Center, Seoul, Republic of Korea; Pasi A. Jänne, M.D., Ph.D, Principal Investigator — Dana-Farber Cancer Institute, Boston, MA, USA
Locations (72):
- United States (15):
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site 2, Los Angeles, California
  - Research Site, Los Angeles, California
  - Research Site, Montebello, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Boca Raton, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Evanston, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Charlotte, North Carolina
  - Research Site, Washington, Washington
- Australia (6):
  - Research Site, Darlinghurst
  - Research site, Fitzroy
  - Research Site, Frankston
  - Research Site, Kogarah
  - Research Site, St Albans
  - Research Site, Woolloongabba
- Research Site, Toronto, Canada
- Germany (5):
  - Research Site, Berlin
  - Research Site, Homburg
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Ulm
- Italy (5):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Rome
- Malaysia (4):
  - Research Site, George Town, Pulau Pinang
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Kuching
- Philippines (5):
  - Research Site, Makati, Kalakhang Maynila
  - Research Site, Pasig, Manila
  - Research Site 2, Manila, National Capital Region
  - Research Site, Manila, National Capital Region
  - Research Site, Cebu
- South Korea (14):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Hwasun
  - Research Site, Incheon
  - Research Site 2, Seongnam-si
  - Research Site, Seongnam-si
  - Research Site 2, Seoul
  - Research Site 3, Seoul
  - Research Site 4, Seoul
  - Research Site 5, Seoul
  - Research Site 6, Seoul
  - Research Site 7, Seoul
  - Research Site 8, Seoul
  - Research Site, Seoul
- Spain (11):
  - Research Site, A Coruña
  - Research Site 2, Barcelona
  - Research Site 3, Barcelona
  - Research Site 4, Barcelona
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site 2, Madrid
  - Research Site, Madrid
  - Research Site, Navarra
  - Research Site 2, Valencia
  - Research Site, Valencia
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site 2, Tainan
  - Research Site, Tainan
  - Research Site 2, Taipei
  - Research Site, Taipei